CLINICAL TRIAL: NCT00070733
Title: The Role of 5-Alpha Reductase in Mediating Testosterone Actions
Brief Title: The Effect of 5-Alpha Reductase on Testosterone in Men
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01HD043348-01 (NIH)
Record Dates: First submitted 2003-10-07; First posted 2003-10-10 (Estimated); Last update posted 2005-11-07 (Estimated); Status verified 2003-10

CONDITIONS: Sex Disorders
Keywords: Testosterone; 5-alpha Reductase; Muscle Strength; Libido; Sexual Function; Muscle Mass; Testosterone 5-alpha-Reductase
MeSH Terms: conditions — Sexual Dysfunction, Physiological | interventions — testosterone enanthate

INTERVENTIONS:
Drug: testosterone enanthate
Drug: duastride

SUMMARY:
The enzyme 5-alpha reductase is present in small amounts in muscle and converts testosterone to dihydrotestosterone (DHT). Testosterone affects lean body tissue, muscle size, muscle strength, and sexual function in men. This study will evaluate how 5-alpha reductase influences the effects of testosterone in young healthy men.

DETAILED DESCRIPTION:
Testosterone, the predominant circulating androgen in men, serves as the active hormone in some target tissues; however, testosterone effects in other target organs require its conversion to two active metabolites, estradiol 17-beta and DHT. The role of 5-alpha reductase in mediating testosterone's effects on muscle and sexual function remains unclear. This study will determine whether 5-alpha reduction of testosterone to DHT is necessary for mediating effects on fat-free mass, muscle size, muscle strength, and leg power in men. The study will also evaluate the necessity of 5-alpha reductase for maintenance of androgen effects on sexual function (sexual desire, overall sexual activity, nocturnal penile tumescence [NPT], response to visual erotic stimulus, and penile rigidity) in men.

Participants in this study will be treated with a drug to suppress endogenous testosterone production. Participants will then be randomly assigned to receive either testosterone and placebo or testosterone and the 5-alpha reductase inhibitor dutasteride. Testosterone will be administered weekly; dutasteride and placebo will both be administered daily. Diet and exercise will be standardized across both groups. Participants will be assessed at study entry and Week 20. Assessments will include measurements such as a DEXA scan, MRI scan, and muscle performance and sexual function tests. Participants will also have blood tests for safety monitoring; blood tests will include measures of hematocrit, liver enzymes (AST and ALT), prostate specific antigen (PSA), and cholesterol.

ELIGIBILITY:
Inclusion Criteria

* General good health and capable of undergoing strength testing
* Normal testosterone (300-1100 ng/dL), LH, and FSH levels

Exclusion Criteria

* Currently participating in competitive sports
* Mental state that would preclude complete understanding of the protocol and compliance
* Disorder known to cause or be associated with hypogonadism (e.g., pituitary tumors, hyperprolactinemia, HIV infection, or Klinefelter's Syndrome)
* More than 20% over ideal body weight
* Disabilities that would prevent participation in strength testing (e.g., amputation of limbs, blindness, severe arthritis, angina, or neurologic disorders such as Parkinson's disease, stroke, or myopathy)
* Uncontrolled hypertension, diabetes, congestive heart failure, or chronic obstructive lung disease
* Alcohol or drug dependence in the 6 months prior to study entry
* Disorders that might be exacerbated by androgen treatment (e.g., benign prostatic hyperplasia or prostate cancer, erythrocytosis [hematocrit > 51% at baseline], or sleep apnea assessed by Berlin's questionnaire)
* Serum PSA levels > 4 microg/L
* AST, ALT, or alkaline phosphatase elevation greater than three times the upper limit of normal
* Creatinine greater than 2 mg/dL
* Medications that might affect muscle or bone metabolism (e.g., glucocorticoid, rhGH, androgenic steroids, oral androgen precursors such as androstenedione or DHEA) or androgen metabolism, action, or clearance (e.g., dilantin, phenobarbitol, aldactone, flutamide, finasteride)

Ages: 21 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 184
Dates: Start 2003-08; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Shalender Bhasin, MD, Principal Investigator — Charles R. Drew University
Locations (1):
- Charles R. Drew University, Los Angeles, California, United States